CLINICAL TRIAL: NCT06393257
Title: Efficacy and Safety of Airway Clearance Technique by Oscillation and Lung Expansion in Patients With Bronchiectasis
Brief Title: Airway Clearance Technique of Oscillation and Lung Expansion in Bronchiectasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230901
Record Dates: First submitted 2024-04-21; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Bronchiectasis Adult
Keywords: bronchiectasis; Airway Clearance Technique
MeSH Terms: conditions — Bronchiectasis | interventions — Drainage, Postural; Expectorants

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of the two groups. No cross-over of the study group will be made
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oscillation and Lung Expansion (Experimental)
  Interventions: Device: Oscillation and Lung Expansion; Drug: Anti-infective therapy; Drug: Mucolytic
- postural drainage (Active Comparator)
  Interventions: Behavioral: Postural drainage; Drug: Anti-infective therapy; Drug: Mucolytic

INTERVENTIONS:
Device: Oscillation and Lung Expansion — A novel airway clearance technology
  Arms: Oscillation and Lung Expansion
Behavioral: Postural drainage — A type of physical therapy used to treat respiratory diseases by changing the patient's body position so that sputum is drained down the respiratory tract so that it can be more easily expelled from the body.
  Arms: postural drainage
Drug: Anti-infective therapy — Antibiotics were used in these patients.
Drug: Mucolytic — Mucolytics were used in these patients.

SUMMARY:
The goal of this prospective randomized controlled trial is to explore the efficacy and safety of Oscillation and Lung Expansion-a airway clearance technology-in bronchiectasis. Participants will receive Oscillation and Lung Expansion or postural drainage randomly in this study. and the symptom, quality of life scores and amount of expectoration will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute exacerbation of bronchiectasis

Exclusion Criteria:

* Haemoptysis greater than 50ml
* state of endangerment
* pneumothorax
* Lung surgery history within 6 months
* Severe heart, brain and nervous system diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
sputum volume in 24h | 2 weeks

SECONDARY OUTCOMES:
Bronchiectasis exacerbation and symptom tool | Assessed at baseline, 2 weeks, 4 weeks, 8 weeks and 12 weeks post-discharge
  BEST score
Quality of life questionnaire-bronchiectasis | Assessed at baseline, 2 weeks, 4 weeks, 8 weeks and 12 weeks post-discharge
  Qol-B score
Leicester Cough Questionnaire | Assessed at baseline, 2 weeks, 4 weeks, 8 weeks and 12 weeks post-discharge
  LCQ score
Bronchiectasis Health Questionnaire | Assessed at baseline, 2 weeks, 4 weeks, 8 weeks and 12 weeks post-discharge
  BHQ score
Time to the first bronchiectasis exacerbation since randomization | Assessed at 4 weeks, 8 weeks and 12 weeks post-discharge
  Time to the first bronchiectasis exacerbation since randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (3):
- China (3):
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai pulmonary hospital, Shanghai, Shanghai Municipality
  - The Shanghai First People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou YM, Wang C, Yao WZ, Chen P, Kang J, Huang SG, Chen BY, Wang CZ, Ni DT, Liu SM, Wang XP, Wang DL, Lu JC, Zheng JP, Zhong NS, Ran PX. [The prevalence and risk factors of bronchiectasis in residents aged 40 years old and above in seven cities in China]. Zhonghua Nei Ke Za Zhi. 2013 May;52(5):379-82. Chinese. PMID 23945301
- [Background] Lin JL, Xu JF, Qu JM. Bronchiectasis in China. Ann Am Thorac Soc. 2016 May;13(5):609-16. doi: 10.1513/AnnalsATS.201511-740PS. PMID 26882271
- [Background] Basavaraj A, Choate R, Addrizzo-Harris D, Aksamit TR, Barker A, Daley CL, Anne Daniels ML, Eden E, DiMango A, Fennelly K, Griffith DE, Johnson MM, Knowles MR, Metersky ML, Noone PG, O'Donnell AE, Olivier KN, Salathe MA, Schmid A, Thomashow B, Tino G, Winthrop KL. Airway Clearance Techniques in Bronchiectasis: Analysis From the United States Bronchiectasis and Non-TB Mycobacteria Research Registry. Chest. 2020 Oct;158(4):1376-1384. doi: 10.1016/j.chest.2020.06.050. Epub 2020 Jul 3. PMID 32622820
- [Background] Munoz G, de Gracia J, Buxo M, Alvarez A, Vendrell M. Long-term benefits of airway clearance in bronchiectasis: a randomised placebo-controlled trial. Eur Respir J. 2018 Jan 11;51(1):1701926. doi: 10.1183/13993003.01926-2017. Print 2018 Jan. PMID 29326318
- [Background] Lee AL, Burge AT, Holland AE. Positive expiratory pressure therapy versus other airway clearance techniques for bronchiectasis. Cochrane Database Syst Rev. 2017 Sep 27;9(9):CD011699. doi: 10.1002/14651858.CD011699.pub2. PMID 28952156
- [Background] Liu Y, Lu HW, Gu SY, Wang WW, Ge J, Jie ZJ, Jia JG, Gao ZT, Li J, Shi JY, Liang S, Cheng KB, Bai JW, Qu JM, Xu JF. Bronchoscopic airway clearance therapy for acute exacerbations of bronchiectasis. EBioMedicine. 2021 Oct;72:103587. doi: 10.1016/j.ebiom.2021.103587. Epub 2021 Sep 16. PMID 34537448
- [Background] Huynh TT, Liesching TN, Cereda M, Lei Y, Frazer MJ, Nahouraii MR, Diette GB. Efficacy of Oscillation and Lung Expansion in Reducing Postoperative Pulmonary Complication. J Am Coll Surg. 2019 Nov;229(5):458-466.e1. doi: 10.1016/j.jamcollsurg.2019.06.004. Epub 2019 Jul 27. PMID 31362061